CLINICAL TRIAL: NCT03055143
Title: A Randomized, Open Label, Two Treatment, Two Period, Two Sequence, Single Dose, Crossover, Bioequivalence Study Of Doxorubicin Hydrochloride Liposome Injection, 2 mg/ml (50 mg/m2 Dose) of Sun Pharma Advanced Research Company Limited, India, And Caelyx® (Doxorubicin Hydrochloride) Liposome Injection, 2 mg/ml (50 mg/m2 Dose) of Schering-Plough, Belgium, in Patients With Metastatic Breast Cancer/Advanced Ovarian Cancer, Under Fed (Normal Breakfast) Conditions.
Brief Title: Study of Doxorubicin in Patients With Metastatic Breast Cancer/Advanced Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: PKD/08/038
Record Dates: First submitted 2017-02-07; First posted 2017-02-16 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer and Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPARC-08-038 (Experimental): 2 mg/ml
  Interventions: Drug: SPARC-08-038; Drug: Ref-08-038
- Ref-08-038 (Active Comparator)
  Interventions: Drug: SPARC-08-038; Drug: Ref-08-038

INTERVENTIONS:
Drug: SPARC-08-038 — 2 mg/ml intravenous infusion
Drug: Ref-08-038 — 2 mg/ml intravenous infusion

SUMMARY:
This was a randomized, multi centre, open label, two treatment, two period, two sequence, single dose, crossover study, with at least 28 days washout between doses, conducted under fed (normal breakfast) conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
2. Patients with metastatic breast cancer/advanced ovarian cancer having age within the range of between 18-55 years.
3. Subjects who had no evidence of underlying disease
4. Subjects who had signed written consent form

Exclusion Criteria:

1. Females who were pregnant, breastfeeding, or are likely to become pregnant
2. Subjects who had any medical condition (except metastatic breast cancer/advanced ovarian cancer) that could jeopardize their health or prejudice the results
3. Subjects deemed uncooperative or noncompliant
4. Smoking or consumption of any nicotine products

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-09-03 (Actual); Primary Completion 2009-11-28 (Actual); Study Completion 2009-11-28 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration | 336 hours

SECONDARY OUTCOMES:
The area under the plasma concentration versus time curve from time 0 to infinity | 336 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhowmik S, Bhowmick S, Maiti K, Chakra A, Shahi P, Jain D, Rajamannar T. Two multicenter Phase I randomized trials to compare the bioequivalence and safety of a generic doxorubicin hydrochloride liposome injection with Doxil(R) or Caelyx(R) in advanced ovarian cancer. Cancer Chemother Pharmacol. 2018 Sep;82(3):521-532. doi: 10.1007/s00280-018-3643-3. Epub 2018 Jul 11. PMID 29995186